CLINICAL TRIAL: NCT01914601
Title: Does King Vision® Videolaryngoscope Reduce Cervical Spine Motion During Endotracheal Intubation? A Cross-over Study.
Brief Title: King Vision and Cervical Spines Movement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KFHU-FBR 0040, MU-R/15.11.04
Record Dates: First submitted 2013-07-28; First posted 2013-08-02 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Need Tracheal Intubation
Keywords: Laryngoscope; Macintosh; King Vision; tracheal intubation; cervical spines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Macintosh-King Vision (Active Comparator): laryngoscopy will be performed with the Macintosh followed by the King Vision laryngoscope
  Interventions: Device: Macintosh-King Vision
- King Vision-Macintosh (Active Comparator): laryngoscopy will be performed with the King Vision followed by the Macintosh laryngoscope.
  Interventions: Device: King Vision-Macintosh

INTERVENTIONS:
Device: Macintosh-King Vision — laryngoscopy will be performed with the Macintosh followed by the King Vision laryngoscope
  Arms: Macintosh-King Vision
Device: King Vision-Macintosh — laryngoscopy will be performed with the King Vision followed by the Macintosh laryngoscope.
  Arms: King Vision-Macintosh

SUMMARY:
Extensive cervical spines movement during endotracheal intubation can result in serious neurological injury, especially in the patients with unrecognized cervical spines injury.[1-2] Moreover, direct laryngoscopy may be difficult if spine movement is limited because of arthritis, disc disease or a small gap between the occiput and the spinous process of the atlas.[3-4]

Video laryngoscopes allow for intubation without alignment of the oral, pharyngeal, and tracheal axes which minimize the cervical movements, especially in the patients with restricted cervical movements. [5,6] Compared with the Macintosh laryngoscope, the use of AirWay Scope decreases median upper cervical-spine movement during intubation under in-line stabilization in patients with normal cervical-spine. [6] Unfortunately, the use video laryngoscopes are associated with longer times to tracheal intubation compared with the traditional techniques which may be attributed to the variable learning curves of the practitioners. [7-9]

The King Vision video laryngoscope® (King Systems Company, a division of Consort Medical, Indianapolis, Indiana, USA) is an anatomically shaped, rigid laryngoscope that uses fiberoptic technology to view the larynx with micro camera offers a 160 degree of view potentially eliminating the need for neck flexion and head extension. [10]

To the best of the authors' knowledge, there is no study has evaluated the King vision laryngoscope regarding the neck movement during routine tracheal intubation under general anesthesia.

DETAILED DESCRIPTION:
Hypothesis:

The investigators hypothesize that the use of King Vision video laryngoscope may reduce the cervical spines movements during endotracheal intubation compared with the Macintosh laryngoscope.

Aim of the study:

The present clinical trial aims to compare the effects of the Macintosh and King Vision laryngoscopes, on cervical spines movement, time to intubation, laryngoscopic view, ease of intubation, number of intubation attempts, and number of optimization maneuvers during tracheal intubation, in the patients undergoing minor elective surgery under propofol-remifentanil-rocuronium anesthesia.

Methods:

Thirty two ASA I-II patients who need tracheal intubation will be included in this randomized cross-over controlled blind comparative study at the author's center after obtaining approval of the local Ethical Committee and an informed written consent from all participants.

The Mallampati airway score, thyromental and sternomental distances, neck extension, and the degree of mouth opening will be evaluated preoperatively as factors predicting difficult intubation.

Sample size calculation:

A priori power analysis of the previous published data [9] showed that the investigators will need to study 14 pairs to detect a 10% difference in the cervical spine extension (occiput-C5) values (25.9 degrees) with a SD of 2.8 degrees, after intubation with of Macintosh laryngoscope, a type-I error of 0.05 and a power of 90%. The investigators will add 10% more patients for a final sample size of 32 patients to account for patients dropping out during the study.

Anesthesia:

Patients will be placed on the operating room table with a rigid board from the shoulders to the occiput with the patient's head rested on a pillow in a position judged by the patient to be neutral. After verification that the patient will be properly centered, the fluoroscopy unit and operating room table will remain fixed for the rest of the study.

Patients' monitoring includes pulse oximetry, noninvasive blood pressure electrocardiography, state and response Entropy (SE and RE) and train of four (TOF)stimulation of the ulnar nerve.

Anesthetic technique will be standardized in all studied. After breathing 100% oxygen for 3 min through a facemask in a neutral position, anesthesia will be induced with fentanyl 2-3µg/kg/min and propofol 2-3 mg/kg to achieve a SE < 50 and the difference between RE and SE less than 10. Rocuronium 0.6 mg.kg will be administered for complete relaxation on the TOF (TOF-GE, Datex-Ohmeda Division, Instrumentarium Corporation, Helsinki, Finland). Anesthesia will be maintained using sevoflurane end-tidal concentrations of 2.5-3.5% in oxygen via a bag-mask for 3 min before endotracheal intubation.

Standard precautions against radiation exposure will be taken, movement of the cervical spines during endotracheal intubation will be studied and recorded with portable X-ray machine. Laryngoscopy will be performed twice, once with the King Vision and once with the Macintosh laryngoscope in random order. For the first device, the patient's mouth will be opened and the tip of the tracheal tube will be introduced into the glottis. The second device will be studied in an identical manner, and intubation will be completed with the second device. The intubators who will participate in the study will receive a standard manikin based training which will be followed with 50 successful endotracheal intubations in the clinical practice with the use of Macintosh and King Vision® laryngoscopes.

The studied data during intubation will be collected by an independent investigator. The intubator will attempt to minimize neck movement during both techniques through the acceptance of the first view [8] that will offer a reasonable opportunity to adequately position the tracheal tube at the glottis opening.

Three lateral radiographs will be taken with a portable X-ray system provides fixed images from which hard copies are generated. Patient will be served as their own control with reference to the first image, which will be obtained after induction of anesthesia before laryngoscopy and intubation, with the patient in neutral position. A further two images, one with the Macintosh and one with King Vision laryngoscopes. These images will be taken at the time of laryngeal exposure, with the tip of the endotracheal tube passing between the vocal cords.

On each image, lines will be drawn to mark the relative position of the occiput, atlas (C1), axis (C2) and the fifth cervical vertebra (C5). The angle between each of these lines will be measured to determine the degree of angulation of C1, C2 and C5 relative to the occiput and each other. [9] The radiographs will be reviewed by a radiology consultant who will be blinded to the order of intubation technique and unfamiliar with the laryngoscopes being used.

Statistical Analysis

Data will be tested for normality using the Kolmogorov-Smirnov test. Fisher exact test will be used for categorical data. Repeated two-way ANOVA and paired t-test will be used to study the changes in the primary and secondary endpoints during each intervention. The Wilcoxon 2 rank sum test will be used for the non-parametric values. The investigators will avoid the carryover effect (persistence of the effect of the first intervention on the operative conditions into the second period) through the comparison of the effects of period (time effect) and the order of treatment using independent t-tests. Data will be expressed as mean ± SD, number (%), or median [range]. A value of P < 0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Sixteen American Society of Anesthesiologists physical status class I-II
* aged 18-65 years
* scheduled for elective minor surgery
* under general anesthesia

Exclusion Criteria:

* predicted or known difficult airway
* history of cervical spine injury
* history of cervical spine surgery
* previous oral surgery
* previous throat surgery
* previous neck surgery
* gastro-esophageal reflux disease
* need for rapid sequence induction
* emergent surgery
* pregnancy
* body mass index higher than 35 kg/m2
* without incisor teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
cervical spine movement | Participants will be followed for the duration of tracheal intubation, an expected average of 60 seconds
  cervical spine movement during tracheal intubation

SECONDARY OUTCOMES:
time to intubation | participants will be followed for the duration of tracheal intubation, an expected average of 60 seconds
  the time when the investigated laryngoscope passes the central incisors to the time when the tip of the tracheal tube passed through the glottis
laryngoscopic view | participants will be followed for the duration of laryngoscopy, an expected average of 90 seconds
  The glottic view during laryngoscopy will be assessed according to the Cormack-Lehane grading system: Grade 1, full view; Grade 2, only arytenoid cartilages visible; Grade 3, only epiglottis visible; and Grade 4, epiglottis not visible
ease of intubation | participants will be followed for the duration of tracheal intubation, an expected average of 60 seconds
  rate the ease of intubation using a 100 mm visual analog scale (0 for much of ease and 100 for extremely difficult).
number of intubation attempts | participants will be followed for the duration of tracheal intubation, an expected average of 60 seconds
number of optimization maneuvers | participants will be followed for the duration of laryngoscopy, an expected average of 90 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Abdulmohsen Al Ghamdi, MD, Principal Investigator — Associate Professor/Chairman of Anesthesiology; Mohamed R El Tahan, MD, Study Director — Associate Professor of Anesthesiology; Alaa M Khidr, MD, Study Chair — Assistant Professor of Anesthesiology; Abdullah s Al Mulhim, MD, Study Chair — Demonstrator of Radiology; Samah A El Kenany, MD, Study Chair — Lecturer of Anesthesiology, Mansoura University, Egypt
Locations (2):
- Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt
- King Fahd Hospital of Dammam University, Khobar, Eastern Province, Saudi Arabia